CLINICAL TRIAL: NCT02161315
Title: A Randomized Study of Steroid Aromatase Inhibitors Versus Progestogens for Non-Steroid Aromatase Inhibitor-resistanced Late Stage Breast Cancer
Brief Title: Steroid Aromatase Inhibitors Versus Progestogens for nSAID-resistanced Late Stage Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CIH-SYH-201205001
Record Dates: First submitted 2014-01-06; First posted 2014-06-11 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2012-02

CONDITIONS: Carcinoma Breast Stage IV
Keywords: SAID, Progestogens, nSAID-resistanced, LSBC
MeSH Terms: conditions — Breast Neoplasms; Simian Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Observation group: Steroid Aromatase Inhibitors
- Control group: Non-Steroid Aromatase Inhibitor

SUMMARY:
Steroid Aromatase Inhibitors and Non-Steroid Aromatase Inhibitors in Late Stage Breast Cancer is the recommended scheme in National Comprehensive Cancer Network (NCCN) guideline. In the past controlled clinical trials with small sample.

DETAILED DESCRIPTION:
A Randomized Study of Steroid Aromatase Inhibitors Versus Progestogens for Non-Steroid Aromatase Inhibitor-resistanced Late Stage Breast Cancer.The primary endpoints of the study is progression free survival (PFS). The secondary endpoints are overall response rate (ORR), overall survival (OS) and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be the postmenopausal women
2. Patients must be diagnosed with advanced breast cancer by imageology，cytology or histopathology
3. Immunohistochemistry shows ER and/or PR positive
4. Patients ECOG score must be 0-2
5. Drug resistant about Non-Steroid Aromatase Inhibitors

Exclusion Criteria:

1. Not suitable for endocrine therapy
2. Have receive the standard Steroid Aromatase Inhibitors treatment
3. Severe hepatic dysfunction

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 80
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
RECIST 1.1 | -7 days

CONTACTS AND LOCATIONS:
Overall Officials: Yehui Shi, M.D., Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China